CLINICAL TRIAL: NCT01722877
Title: Safety and Effectiveness of JetStream (JS) Atherectomy in Femoropopliteal In-Stent Restenotic Lesions: A Prospective Registry
Brief Title: JetStream (JS) Atherectomy in Femoropopliteal In-Stent Restenotic Lesions
Acronym: JetStreamISR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Midwest Cardiovascular Research Foundation (Other)
Collaborators: MEDRAD, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JS-ISR-001, version 1, Rev 2
Record Dates: First submitted 2012-11-05; First posted 2012-11-07 (Estimated); Results first posted 2017-05-05 (Actual); Last update posted 2020-03-03 (Actual); Status verified 2020-02

CONDITIONS: Restenosis; Peripheral Vascular Disease
Keywords: Restenosis; aspiration; in-stent restenosis; atherectomy; superficial femoral artery; popliteal artery
MeSH Terms: conditions — Peripheral Vascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- JetStream Atherectomy (Experimental): Jetstream NAVITUS System is a rotating, aspirating, expandable catheter for active removal of atherosclerotic disease and thrombus in peripheral vasculature.
  Interventions: Device: JetStream Navitus

INTERVENTIONS:
Device: JetStream Navitus — Study to use Jetstream device for use of in-stent restenosis in femoral popliteal artery.

SUMMARY:
Several studies have shown that stenting of the femoropopliteal artery in the lower leg leads to improved overall results compared to balloon angioplasty alone. However, scar tissue development can occur within the stent, a process called restenosis. Treatment of these in-stent restenotic lesions has a high procedural success rate but recurrence of scar tissue is frequently seen. Several methods have been proposed to treat in-stent restenosis in the lower leg arteries but mixed results have been noted. In this study we hypothesize that simultaneous tissue excision and aspiration using the JetStream Navitus device (Medrad) can lead to a high rate of acute procedural success with low intraprocedural complications and an acceptable recurrence rate of restenosis at 6-month follow-up.

DETAILED DESCRIPTION:
Data not available yet.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is 18 years of age or older.
2. Subject presents with clinical evidence of peripheral arterial disease with ISR in the femoropopliteal segment (includes common femoral, superficial femoral and popliteal)
3. Subject presents with a Rutherford Classification of 1-5 and has symptoms of rest limb pain, ulcerations or claudication.
4. Target lesion(s) must be viewed angiographically and have ≥50% stenosis.
5. The atherectomy wire must be placed entirely across all lesions to be treated with no visible evidence of clear or suspected subintimal/substent wire passage.
6. The main target vessel reference diameter must be at least 5 mm.
7. One patent distal run-off vessel with brisk flow is required.
8. Patient is an acceptable candidate for percutaneous intervention using the Jetstream NAVITUS System in accordance with its labeled instructions for use.
9. Patient has signed approved informed consent.
10. Patient is willing to comply with the follow-up evaluations at specified times.

Exclusion Criteria:

1. Subject is unable to understand the study or has a history of non-compliance with medical advice.
2. Subject is unwilling or unable to sign the Informed Consent Form (ICF).
3. Subject is currently enrolled in another clinical investigational study that might clinically interfere with the current study endpoints (e.g., limit use of study-recommended medications, etc.).
4. Subject is pregnant or planning to become pregnant within the study period.
5. Subject has a known sensitivity to contrast media and the sensitivity cannot be adequately pre-medicated for.
6. Subject is diagnosed with chronic renal failure or has a creatinine level > 2.5 mg/dl and is not on chronic dialysis.
7. Subject has a known allergy to heparin, ASA, Plavix.
8. Subject has a history of bleeding disorders or platelet count < 80,000 cells/ml.
9. Subject experiences ongoing cardiac problems (e.g., cardiac arrhythmias, congestive heart failure exacerbation, myocardial infarction, etc.) that, per the investigator, would not make the subject an ideal candidate for study procedures.
10. Subject has a CVA or TIA within 4 weeks prior to JetStream procedure.
11. Subject has an anticipated life span of less than 6 months.
12. Subject is suspected of having an active systemic infection.
13. Subject per the investigator's medical judgment must be excluded from the study.
14. Limited vascular access that precludes safe advancement of the Jetstream NAVITUS System to the target lesion(s).
15. Patient has evidence of intracranial or gastrointestinal bleeding within the past 3 months.
16. Patient has had severe trauma, fracture, major surgery or biopsy of a parenchymal organ within the past 14 days.
17. Patient has any planned surgical intervention or endovascular procedure within 15 days after the index procedure.
18. Use of another debulking device during the index procedure prior to the Jetstream NAVITUS System.
19. Use of another debulking device after the Jetstream NAVITUS system.

    -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2012-10; Primary Completion 2014-08 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas W Shammas, MD, MS, Principal Investigator — Midwest Cardiovascular Research Foundation
Locations (2):
- United States (2):
  - Trinity Bettendorf Medical Center, Bettendorf, Iowa
  - VA Medical Center, Dallas, Texas

IPD SHARING:
Plan to Share IPD: Yes
Manuscript will be published in JEVT early 2016

REFERENCES:
- [Derived] Shammas NW, Shammas GA, Banerjee S, Popma JJ, Mohammad A, Jerin M. JetStream Rotational and Aspiration Atherectomy in Treating In-Stent Restenosis of the Femoropopliteal Arteries: Results of the JETSTREAM-ISR Feasibility Study. J Endovasc Ther. 2016 Apr;23(2):339-46. doi: 10.1177/1526602816634028. Epub 2016 Feb 26. PMID 26921281

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 29 patients with FP ISR in 32 limbs were treated at 2 medical centers by 2 operators from October 2012 to August 2014. Patients were eligible only if they had a more or equal 50% in-stent restenotic lesion in the superficial femoral or popliteal arteries (estimated diameter ≥5 mm), Rutherford category 1-5, and at least one patent runoff vessel.
Pre-assignment Details: Patients were excluded if they were not able to give informed consent, had a creatinine level >2.5 mg/dL, were unable to take antiplatelet drugs, or had a planned surgical or endovascular procedure within 15 days of the index procedure. After consenting, patient were excluded if had denovo disease or no in-stent restenosis in the target vessel.
Units Other Than Participants: limbs
Groups:
- JetStream Atherectomy: Jetstream NAVITUS System is a rotating, aspirating, expandable catheter for active removal of atherosclerotic disease and thrombus in peripheral vasculature. In this study, Jetstream Navitus was used to treat in-stent restenosis in femoral popliteal artery.
Period: Overall Study
Arm/Group | JetStream Atherectomy
Started | 29; 32 limbs
Completed | 27; 29 limbs
Not Completed | 2; 3 limbs
Not completed — Death | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Groups:
- JetStream Atherectomy: Jetstream NAVITUS System is a rotating, aspirating, expandable catheter for active removal of atherosclerotic disease and thrombus in peripheral vasculature. In this study, Jetstream Navitus was used to treat in-stent restenosis in femoral popliteal artery. Patients were eligible for the study only if they had a more or equal 50% in-stent restenotic lesion in the superficial femoral or popliteal arteries (estimated diameter ≥5 mm), Rutherford category 1-5 ischemia, and at least one patent infrapopliteal runoff vessel. Patients were excluded if they were not able to give informed consent, had a creatinine level >2.5 mg/dL, were unable to take antiplatelet drugs, or had a planned surgical or endovascular procedure within 15 days of the index procedure.The JetStream was used as a first modality of treatment, no other debulking devices, cutting/scoring balloons, or cryogenic balloons were allowed.
Arm/Group | JetStream Atherectomy
Number analyzed (Participants) | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.9 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 11
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 29

OUTCOME MEASURES:

1. Primary Outcome: Acute Procedural Success
Description: Acute procedural success is defined as less than or equal to 30 percent residual stenosis (via Quantitative Vascular Analysis) at the index lesion post JestStream atherectomy and final adjunctive treatment And with no serious adverse events.
Time Frame: intraprocedural
Measure: Count of Units; unit: limbs
Units Other Than Participants: limbs
Arm/Group | JetStream Atherectomy
Number analyzed (Participants) | 29
Number analyzed (limbs) | 32
limbs | 29

2. Secondary Outcome: Patency
Description: Patency is defined as Peak Systolic Velocity Ratio (PSVR) of < 2.4 by duplex criteria. PSVR is obtained by dividing velocity (cm/sec) at the lesion site to the velocity immediately proximal to the lesion.
Time Frame: 6 months
Population: Only 25 limbs had duplex ultrasound at 6 months.
Measure: Number; unit: Percentage of patent limbs
Units Other Than Participants: limbs
Groups:
- JetStream Atherectomy: Jetstream NAVITUS System is a rotating, aspirating, expandable catheter for active removal of atherosclerotic disease and thrombus in peripheral vasculature. In this study, Jetstream Navitus was used to treat in-stent restenosis in femoral popliteal artery.
  25 patients in the Jetstream ISR study had a duplex Ultrasound to evaluate for patency of treated vessel at 6 months. Remaining patients did not have a DUS.
Arm/Group | JetStream Atherectomy
Number analyzed (Participants) | 25
Number analyzed (limbs) | 25
Percentage of patent limbs | 72

3. Secondary Outcome: Target Lesion Revascularization
Description: Reintervention on the same index lesion at 6 months
Time Frame: 6 months
Measure: Count of Units; unit: lesions
Units Other Than Participants: lesions
Arm/Group | JetStream Atherectomy
Number analyzed (Participants) | 29
Number analyzed (lesions) | 29
lesions | 4

4. Other Pre Specified Outcome: Acute Device Success
Description: Acute device success is defined as less than or equal to 50% residual stenosis at the index lesion using the JetStream device alone and with no adjunctive balloon angioplasty therapy (via Quantitative Vascular Analysis) and with no serious adverse events.
Time Frame: intraprocedural
Measure: Count of Units; unit: limbs
Units Other Than Participants: limbs
Arm/Group | JetStream Atherectomy
Number analyzed (Participants) | 29
Number analyzed (limbs) | 29
limbs | 22

ADVERSE EVENTS:
Time Frame: 6 months
Description: Death
Arm/Group | JetStream Atherectomy
All-Cause Mortality (participants affected / at risk) | 1/29
Serious Adverse Events (participants affected / at risk) | 4/29
Other Adverse Events (participants affected / at risk) | 3/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | JetStream Atherectomy (N=29)
Target lesion revascularization (Vascular disorders) | 4 (4) — retreatment of the same lesion at 6 month
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | JetStream Atherectomy (N=29)
non target vessel revascularization (Vascular disorders) | 3 (3) — treatment of a non target vessel
COPD exacerbation (Respiratory, thoracic and mediastinal disorders) | 2 (2) — worsening chronic obstructive pulmonary disease symptoms

LIMITATIONS AND CAVEATS:
This is a feasibility study that will need to be validated with larger multicenter trials.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No